CLINICAL TRIAL: NCT03823378
Title: A Phase 2, Multicenter, Double-Blind, Parallel Group Long Term Extension Study in Rheumatoid Arthritis Subjects Who Have Completed a Preceding Phase 2 Randomized Controlled Trial With ABBV-105 Given Alone or in Combination With Upadacitinib (ABBV-599)
Brief Title: A Study in Rheumatoid Arthritis Patients Who Have Completed a Preceding Study With ABBV-105 Given Alone or in Combination With Upadacitinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study M16-763 was terminated early as the benefit of each treatment arm from the feeder study (Study M16-063) did not provide appreciable evidence of differentiated clinical effect to warrant further long-term continuation.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-763; 2018-002306-31 (EudraCT Number)
Record Dates: First submitted 2019-01-08; First posted 2019-01-30 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Elsubrutinib; ABBV-105; Upadacitinib; ABBV-599; Rheumatoid Arthritis (RA); Long-term extension (LTE)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- ABBV-599 in M16-063/ABBV-599 in M16-763 (Experimental): 60 mg elsubrutinib capsule once a day by mouth for 48 weeks; 15 mg film-coated upadacitinib tablet once a day by mouth for 48 weeks
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- ABBV-105 60 mg/UPA placebo (Experimental): 60 mg elsubrutinib capsule once a day by mouth for 48 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 48 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- ABBV-105 20 mg/UPA placebo (Experimental): 20 mg elsubrutinib capsule once a day by mouth for 48 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 48 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- ABBV-105 5 mg/UPA placebo (Experimental): 5 mg elsubrutinib capsule once a day by mouth for 48 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 48 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- UPA 15 mg/ABBV-105 placebo (Experimental): 15 mg film-coated upadacitinib tablet once a day by mouth for 48 weeks; placebo capsule for elsubrutinib once a day by mouth for 48 weeks
  Interventions: Drug: Upadacitinib; Drug: Placebo for elsubrutinib
- Placebo in M16-063/ABBV-599 in M16-763 (Experimental): Placebo in M16-063; 60 mg elsubrutinib capsule once a day by mouth for 48 weeks and 15 mg film-coated upadacitinib tablet once a day by mouth for 48 weeks in M16-763
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib

INTERVENTIONS:
Drug: Elsubrutinib — Elsubrutinib capsule will be administered orally.
  Other Names: ABBV-105
  Arms: ABBV-105 20 mg/UPA placebo; ABBV-105 5 mg/UPA placebo; ABBV-105 60 mg/UPA placebo; ABBV-599 in M16-063/ABBV-599 in M16-763; Placebo in M16-063/ABBV-599 in M16-763
Drug: Upadacitinib — Upadacitinib tablet will be administered orally.
  Other Names: ABT-494
  Arms: ABBV-599 in M16-063/ABBV-599 in M16-763; Placebo in M16-063/ABBV-599 in M16-763; UPA 15 mg/ABBV-105 placebo
Drug: Placebo for elsubrutinib — Placebo capsule for elsubrutinib will be administered orally.
  Arms: UPA 15 mg/ABBV-105 placebo
Drug: Placebo for upadacitinib — Upadacitinib placebo tablet will be administered orally.
  Arms: ABBV-105 20 mg/UPA placebo; ABBV-105 5 mg/UPA placebo; ABBV-105 60 mg/UPA placebo

SUMMARY:
This was a long-term extension (LTE) study to assess the safety, tolerability, and efficacy of ABBV-105 (elsubrutinib [ELS]) and ABBV-599 (ELS 60 mg and upadacitinib [UPA] 15 mg) in participants with rheumatoid arthritis (RA) who completed Study M16-063 (NCT03682705).

DETAILED DESCRIPTION:
This was a Phase 2, double-blind, multicenter, long-term extension (LTE) study to assess the safety, tolerability, and efficacy of 3 doses of ABBV-105 (elsubrutinib [ELS] 5 mg, 20 mg, and 60 mg) and ABBV-599 (ELS 60 mg and upadacitinib [UPA] 15 mg) in adults with active rheumatoid arthritis with inadequate response or intolerance to biologic disease-modifying antirheumatic drugs (bDMARDs). Participants who successfully completed treatment in the feeder Study M16-063, a Phase 2 dose exploratory study, were eligible to participate in this study. Those who met eligibility criteria and entered this study receiving ELS, ABBV-599, or UPA from Study M16-063 continued on their previously assigned treatment through termination of this study. Participants originally randomized to placebo in Study M16-063 rolled over to ABBV-599 in a blinded fashion in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed Study M16-063
* Participant has not developed any laboratory or clinical discontinuation criteria as defined in the Study M16-063 protocol
* Participant is willing and/or able to comply with procedures required in the current study protocol

Exclusion Criteria:

* Participant is currently enrolled or planning to enroll in another interventional clinical study while participating in this study (except the preceding study M16-063)
* Participant requires vaccination with any live vaccine during study participation, including at least 30 days after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (30):
- Belgium (2):
  - Cliniques Universitaires Saint Luc /ID# 207719, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Leuven /ID# 207722, Leuven
- Canada (5):
  - Rheumatology Research Assoc /ID# 207769, Edmonton, Alberta
  - Manitoba Clinic /ID# 206852, Winnipeg, Manitoba
  - CIADS Research Co Ltd /ID# 206853, Winnipeg, Manitoba
  - Mount Sinai Hosp.-Toronto /ID# 206851, Toronto, Ontario
  - Dr. Latha Naik /ID# 213440, Saskatoon, Saskatchewan
- Czechia (4):
  - Revmatolog s.r.o. /ID# 209941, Jihlava, Jihlava
  - Revmatologicky ustav Praha /ID# 209943, Prague, Praha 2
  - Revmatologie MUDr. Klara Sirova /ID# 209944, Ostrava
  - CCR Czech a.s /ID# 209942, Pardubice
- Hungary (5):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 208186, Miskolc, Borsod-Abauj Zemplen county
  - Szabolcs-Szatmar-Bereg Megyei Korhazak & Egyetemi Oktatokorhaz /ID# 208184, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Revita Reumatologiai Rendelo /ID# 208187, Budapest
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 208188, Székesfehérvár
  - Vital Medical Center Orvosi-es Fogaszati Kozpont /ID# 208185, Veszprém
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 209902, Krakow, Lesser Poland Voivodeship
  - McBk Sc /Id# 212577, Grodzisk Mazowiecki, Masovian Voivodeship
  - NBR Polska /ID# 209904, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j. /ID# 212578, Bialystok, Podlaskie Voivodeship
  - Reumatika - Centrum Reumatologii NZOZ /ID# 209903, Warsaw
- Spain (8):
  - Hospital Universitario A Coruña - CHUAC /ID# 207732, A Coruña, A Coruna
  - Hospital Unversitario Marques de Valdecilla /ID# 207729, Santander, Cantabria
  - Hospital Regional de Malaga /ID# 207735, Málaga, Malaga
  - Hospital Clinic /ID# 207740, Barcelona
  - Hospital Universitario Basurto /ID# 207737, Bilbao
  - Hospital Universitario Virgen de las Nieves /ID# 209975, Granada
  - Hospital Clinico Universitario San Carlos /ID# 207738, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 207739, Valencia
- University of Oxford /ID# 210571, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants
Period: Overall Study
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Started | 28 | 16 | 12 | 12 | 20 | 9
Completed | 7 | 0 | 2 | 2 | 2 | 1
Not Completed | 21 | 16 | 10 | 10 | 18 | 8
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 2 | 0 | 1
Not completed — Other, not specified | 19 | 12 | 6 | 8 | 17 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who completed Study M16-063 and received at least 1 dose of assigned study drug in Study M16-763
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763 | Total
Number analyzed (Participants) | 28 | 16 | 12 | 12 | 20 | 9 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.64) | 58.6 (8.75) | 58.5 (12.07) | 54.5 (12.21) | 61.7 (8.99) | 59.4 (9.48) | 58.5 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 12 | 8 | 18 | 7 | 77
  Male | 10 | 2 | 0 | 4 | 2 | 2 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 15 | 12 | 12 | 20 | 9 | 95
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
Duration of Rheumatoid Arthritis Diagnosis [Mean (Standard Deviation); unit: years] | 10.024 (5.6087) | 14.212 (9.0327) | 5.435 (3.2458) | 9.466 (6.6508) | 13.571 (7.8086) | 9.684 (5.6087) | 10.778 (7.0861)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either having a reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Time Frame: On or after the first dose of study drug in Study M16-763, and up to 30 days after the last dose of study drug in Study M16-763, up to 52 weeks
Population: Safety Analysis Set: all participants who completed Study M16-063 and received at least 1 dose of assigned study drug in Study M16-763
Measure: Count of Participants; unit: Participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 28 | 16 | 12 | 12 | 20 | 9
Participants | 11 | 10 | 3 | 5 | 7 | 3

2. Secondary Outcome: Change in Disease Activity Score 28 C-reactive Protein (DAS28-CRP) From Baseline of Study M16-063 at Each Study Visit in Study M16-763
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: Full Analysis Set: all participants who completed Study M16-063 and received at least 1 dose of assigned study drug in Study M16-763 with available data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 7 | 10 | 18 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 10 | 18 | 8
  Week 18 | -3.27 [-3.79 to -2.75] | -1.98 [-2.83 to -1.12] | -1.93 [-3.01 to -0.85] | -2.55 [-3.50 to -1.60] | -3.88 [-4.63 to -3.14] | -2.87 [-4.05 to -1.68]
  Week 24: number analyzed (Participants) | 26 | 13 | 7 | 10 | 17 | 7
  Week 24 | -3.43 [-3.90 to -2.95] | -2.62 [-3.56 to -1.68] | -2.02 [-3.18 to -0.86] | -3.20 [-4.10 to -2.30] | -4.02 [-4.62 to -3.43] | -3.61 [-4.94 to -2.28]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 10 | 16 | 8
  Week 30 | -3.17 [-3.86 to -2.47] | -2.37 [-3.71 to -1.03] | -1.45 [-2.30 to -0.60] | -3.30 [-4.43 to -2.17] | -3.84 [-4.56 to -3.12] | -4.08 [-4.73 to -3.44]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 10 | 12 | 6
  Week 36 | -3.45 [-4.14 to -2.77] | -3.12 [-3.99 to -2.25] | -1.63 [-2.37 to -0.89] | -3.00 [-4.17 to -1.83] | -4.15 [-5.02 to -3.29] | -3.77 [-4.79 to -2.74]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 8 | 8 | 6
  Week 48 | -3.55 [-4.32 to -2.78] | -2.77 [-4.92 to -0.62] | -1.68 [-3.10 to -0.27] | -3.16 [-4.49 to -1.84] | -4.38 [-5.67 to -3.09] | -3.86 [-4.88 to -2.85]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -4.06 [-4.88 to -3.25] | -3.21 [-22.18 to 15.75] | -2.55 [-6.90 to 1.79] | -3.41 [-4.92 to -1.89] | -4.12 [-5.43 to -2.81] | -3.69 [-5.19 to -2.19]

3. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Disease Activity Score 28 C-reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Low Disease Activity (LDA) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than or equal to 3.2.
Time Frame: Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 27 | 15 | 9 | 10 | 18 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 23 | 15 | 9 | 10 | 18 | 8
  Week 18 | 78.3 [58.10 to 90.34] | 26.7 [10.90 to 51.95] | 44.4 [18.88 to 73.33] | 20.0 [5.67 to 50.98] | 77.8 [54.79 to 91.00] | 62.5 [30.57 to 86.32]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 7
  Week 24 | 77.8 [59.24 to 89.39] | 53.8 [29.14 to 76.79] | 44.4 [18.88 to 73.33] | 50.0 [23.66 to 76.34] | 88.2 [65.66 to 96.71] | 85.7 [48.69 to 97.43]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | 78.3 [58.10 to 90.34] | 76.9 [49.74 to 91.82] | 28.6 [8.22 to 64.11] | 60.0 [31.27 to 83.18] | 87.5 [63.98 to 96.50] | 100 [67.56 to 100.00]
  Week 36: number analyzed (Participants) | 24 | 8 | 4 | 10 | 12 | 6
  Week 36 | 87.5 [69.00 to 95.66] | 87.5 [52.91 to 97.76] | 25.0 [4.56 to 69.94] | 40.0 [16.82 to 68.73] | 91.7 [64.61 to 98.51] | 100 [60.97 to 100.00]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 6
  Week 48 | 77.8 [54.79 to 91.00] | 66.7 [30.00 to 90.32] | 50.0 [15.00 to 85.00] | 37.5 [13.68 to 69.43] | 87.5 [52.91 to 97.76] | 100 [60.97 to 100.00]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | 100 [70.09 to 100.00] | 50.0 [9.45 to 90.55] | 100 [34.24 to 100.00] | 60.0 [23.07 to 88.24] | 100 [56.55 to 100.00] | 75.0 [30.06 to 95.44]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Disease Activity Score 28 C-reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Clinical Remission (CR) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than 2.6.
Time Frame: Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 27 | 15 | 9 | 10 | 18 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 23 | 15 | 9 | 10 | 18 | 8
  Week 18 | 56.5 [36.81 to 74.37] | 20.0 [7.05 to 45.19] | 11.1 [1.99 to 43.50] | 20.0 [5.67 to 50.98] | 77.8 [54.79 to 91.00] | 50.0 [21.52 to 78.48]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 7
  Week 24 | 70.4 [51.52 to 84.15] | 53.8 [29.14 to 76.79] | 33.3 [12.06 to 64.58] | 30.0 [10.78 to 60.32] | 70.6 [46.87 to 86.72] | 71.4 [35.89 to 91.78]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | 65.2 [44.89 to 81.19] | 46.2 [23.21 to 70.86] | 0 [0.00 to 35.43] | 40.0 [16.82 to 68.73] | 87.5 [63.98 to 96.50] | 100 [67.56 to 100.00]
  Week 36: number analyzed (Participants) | 24 | 8 | 4 | 10 | 12 | 6
  Week 36 | 66.7 [46.71 to 82.03] | 62.5 [30.57 to 86.32] | 0 [0.00 to 48.99] | 20.0 [5.67 to 50.98] | 75.0 [46.77 to 91.11] | 66.7 [30.00 to 90.32]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 6
  Week 48 | 72.2 [49.13 to 87.50] | 66.7 [30.00 to 90.32] | 0 [0.00 to 48.99] | 25.0 [7.15 to 59.07] | 62.5 [30.57 to 86.32] | 83.3 [43.65 to 96.99]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | 77.8 [45.26 to 93.68] | 50.0 [9.45 to 90.55] | 50.0 [9.45 to 90.55] | 0 [0.00 to 43.45] | 60.0 [23.07 to 88.24] | 75.0 [30.06 to 95.44]

5. Secondary Outcome: Change in Clinical Disease Activity Index (CDAI) From Baseline of Study M16-063
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 7 | 9 | 17 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 7 | 17 | 8
  Week 18 | -33.68 [-40.72 to -26.64] | -23.77 [-32.65 to -14.90] | -19.16 [-28.05 to -10.26] | -27.00 [-42.89 to -11.11] | -36.01 [-44.11 to -27.91] | -28.65 [-37.00 to -20.30]
  Week 24: number analyzed (Participants) | 26 | 13 | 7 | 9 | 16 | 8
  Week 24 | -33.47 [-39.66 to -27.27] | -27.20 [-34.18 to -20.22] | -19.84 [-30.65 to -9.03] | -35.59 [-45.25 to -25.93] | -38.27 [-45.66 to -30.88] | -32.93 [-41.70 to -24.15]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 9 | 15 | 8
  Week 30 | -32.07 [-40.11 to -24.03] | -22.40 [-34.25 to -10.55] | -16.72 [-22.28 to -11.16] | -35.92 [-46.64 to -25.20] | -36.86 [-46.20 to -27.52] | -34.00 [-42.21 to -25.79]
  Week 36: number analyzed (Participants) | 21 | 8 | 3 | 9 | 11 | 6
  Week 36 | -35.28 [-43.23 to -27.33] | -28.86 [-36.56 to -21.16] | -19.17 [-32.10 to -6.23] | -33.99 [-47.10 to -20.88] | -42.20 [-52.14 to -32.26] | -32.92 [-41.43 to -24.40]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 7 | 8 | 5
  Week 48 | -36.26 [-45.44 to -27.08] | -22.58 [-41.15 to -4.02] | -18.87 [-36.40 to -1.33] | -34.77 [-49.11 to -20.44] | -45.69 [-57.45 to -33.93] | -35.72 [-45.75 to -25.69]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 4 | 5 | 4
  Week 60 | -37.99 [-49.56 to -26.41] | -29.70 [-216.48 to 157.08] | -24.95 [-78.95 to 29.05] | -37.20 [-56.11 to -18.29] | -43.98 [-58.77 to -29.19] | -34.38 [-46.14 to -22.61]

6. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Clinical Disease Activity Index (CDAI) Criteria
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. Low Disease Activity (LDA) based on CDAI is defined as achieving a total CDAI score of less than or equal to 10.
Time Frame: Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 27 | 15 | 9 | 10 | 18 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 23 | 15 | 9 | 8 | 18 | 8
  Week 18 | 82.6 [62.86 to 93.02] | 40.0 [19.82 to 64.25] | 44.4 [18.88 to 73.33] | 50.0 [21.52 to 78.48] | 77.8 [54.79 to 91.00] | 62.5 [30.57 to 86.32]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 8
  Week 24 | 88.9 [71.94 to 96.15] | 69.2 [42.37 to 87.32] | 55.6 [26.67 to 81.12] | 80.0 [49.02 to 94.33] | 88.2 [65.66 to 96.71] | 100 [67.56 to 100.00]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | 78.3 [58.10 to 90.34] | 76.9 [49.74 to 91.82] | 42.9 [15.82 to 74.95] | 80.0 [49.02 to 94.33] | 81.3 [56.99 to 93.41] | 100 [67.56 to 100.00]
  Week 36: number analyzed (Participants) | 22 | 8 | 4 | 10 | 12 | 6
  Week 36 | 86.4 [66.67 to 95.25] | 87.5 [52.91 to 97.76] | 75.0 [30.06 to 95.44] | 70.0 [39.68 to 89.22] | 83.3 [55.20 to 95.30] | 100 [60.97 to 100.00]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 5
  Week 48 | 77.8 [54.79 to 91.00] | 66.7 [30.00 to 90.32] | 75.0 [30.06 to 95.44] | 62.5 [30.57 to 86.32] | 87.5 [52.91 to 97.76] | 100 [56.55 to 100.00]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | 100 [70.09 to 100.00] | 50.0 [9.45 to 90.55] | 100 [34.24 to 100.00] | 80.0 [37.55 to 96.38] | 80.0 [37.55 to 96.38] | 75.0 [30.06 to 95.44]

7. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Clinical Disease Activity Index (CDAI) Criteria
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. Complete Remission (CR) based on CDAI is defined as achieving a total CDAI score of less than or equal to 2.8.
Time Frame: Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 27 | 15 | 9 | 10 | 18 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 23 | 15 | 9 | 8 | 18 | 8
  Week 18 | 17.4 [6.98 to 37.14] | 13.3 [3.74 to 37.88] | 11.1 [1.99 to 43.50] | 12.5 [2.24 to 47.09] | 55.6 [33.72 to 75.44] | 25.0 [7.15 to 59.07]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 8
  Week 24 | 29.6 [15.85 to 48.48] | 23.1 [8.18 to 50.26] | 11.1 [1.99 to 43.50] | 10.0 [1.79 to 40.42] | 58.8 [36.01 to 78.39] | 50.0 [21.52 to 78.48]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | 26.1 [12.55 to 46.47] | 30.8 [12.68 to 57.63] | 14.3 [2.57 to 51.31] | 30.0 [10.78 to 60.32] | 43.8 [23.10 to 66.82] | 87.5 [52.91 to 97.76]
  Week 36: number analyzed (Participants) | 22 | 8 | 4 | 10 | 12 | 6
  Week 36 | 36.4 [19.73 to 57.05] | 25.0 [7.15 to 59.07] | 25.0 [4.56 to 69.94] | 10.0 [1.79 to 40.42] | 41.7 [19.33 to 68.05] | 50.0 [18.76 to 81.24]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 5
  Week 48 | 44.4 [24.56 to 66.28] | 33.3 [9.68 to 70.00] | 0 [0.00 to 48.99] | 12.5 [2.24 to 47.09] | 50.0 [21.52 to 78.48] | 100 [56.55 to 100.00]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | 33.3 [12.06 to 64.58] | 50.0 [9.45 to 90.55] | 50.0 [9.45 to 90.55] | 20.0 [3.62 to 62.45] | 60.0 [23.07 to 88.24] | 50.0 [15.00 to 85.00]

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: Participants who met the following 3 conditions for improvement from baseline of Study M16-063 were classified as meeting the American College of Rheumatology 20% response (ACR20) criteria:
  1. ≥ 20% improvement in 68-tender joint count from Baseline of Study M16-063
  2. ≥ 20% improvement in 66-swollen joint count from Baseline of Study M16-063 and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters from Baseline of Study M16-063:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 7 | 10 | 17 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 9 | 17 | 8
  Week 18 | 90.9 [72.19 to 97.47] | 80.0 [54.81 to 92.95] | 57.1 [25.05 to 84.18] | 66.7 [35.42 to 87.94] | 88.2 [65.66 to 96.71] | 75.0 [40.93 to 92.85]
  Week 24: number analyzed (Participants) | 26 | 14 | 7 | 9 | 16 | 8
  Week 24 | 96.2 [81.11 to 99.32] | 92.9 [68.53 to 98.73] | 85.7 [48.69 to 97.43] | 77.8 [45.26 to 93.68] | 93.8 [71.67 to 98.89] | 100 [67.56 to 100.00]
  Week 30: number analyzed (Participants) | 22 | 13 | 6 | 10 | 16 | 8
  Week 30 | 86.4 [66.67 to 95.25] | 69.2 [42.37 to 87.32] | 50.0 [18.76 to 81.24] | 80.0 [49.02 to 94.33] | 87.5 [63.98 to 96.50] | 100 [67.56 to 100.00]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 9 | 12 | 6
  Week 36 | 87.0 [67.87 to 95.46] | 87.5 [52.91 to 97.76] | 66.7 [20.77 to 93.85] | 88.9 [56.50 to 98.01] | 91.7 [64.61 to 98.51] | 83.3 [43.65 to 96.99]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 7 | 8 | 6
  Week 48 | 94.1 [73.02 to 98.95] | 83.3 [43.65 to 96.99] | 66.7 [20.77 to 93.85] | 85.7 [48.69 to 97.43] | 87.5 [52.91 to 97.76] | 100 [60.97 to 100.00]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 4 | 5 | 4
  Week 60 | 88.9 [56.50 to 98.01] | 100 [34.24 to 100.00] | 100 [34.24 to 100.00] | 75.0 [30.06 to 95.44] | 100 [56.55 to 100.00] | 100 [51.01 to 100.00]

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: Participants who met the following 3 conditions for improvement from baseline of Study M16-063 were classified as meeting the American College of Rheumatology 50% response (ACR50) criteria:
  1. ≥ 50% improvement in 68-tender joint count from Baseline of Study M16-063
  2. ≥ 50% improvement in 66-swollen joint count from Baseline of Study M16-063 and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters from Baseline of Study M16-063:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 10 | 10 | 17 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 22 | 15 | 10 | 10 | 17 | 8
  Week 18 | 68.2 [47.32 to 83.64] | 46.7 [24.81 to 69.88] | 40.0 [16.82 to 68.73] | 40.0 [16.82 to 68.73] | 70.6 [46.87 to 86.72] | 62.5 [30.57 to 86.32]
  Week 24: number analyzed (Participants) | 26 | 14 | 7 | 9 | 16 | 8
  Week 24 | 76.9 [57.95 to 88.97] | 64.3 [38.76 to 83.66] | 42.9 [15.82 to 74.95] | 66.7 [35.42 to 87.94] | 87.5 [63.98 to 96.50] | 100 [67.56 to 100.00]
  Week 30: number analyzed (Participants) | 22 | 13 | 6 | 10 | 16 | 8
  Week 30 | 63.6 [42.95 to 80.27] | 61.5 [35.52 to 82.29] | 16.7 [3.01 to 56.35] | 60.0 [31.27 to 83.18] | 87.5 [63.98 to 96.50] | 100 [67.56 to 100.00]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 9 | 12 | 6
  Week 36 | 82.6 [62.86 to 93.02] | 62.5 [30.57 to 86.32] | 33.3 [6.15 to 79.23] | 66.7 [35.42 to 87.94] | 75.0 [46.77 to 91.11] | 66.7 [30.00 to 90.32]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 7 | 8 | 6
  Week 48 | 82.4 [58.97 to 93.81] | 66.7 [30.00 to 90.32] | 66.7 [20.77 to 93.85] | 71.4 [35.89 to 91.78] | 87.5 [52.91 to 97.76] | 83.3 [43.65 to 96.99]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 4 | 5 | 4
  Week 60 | 88.9 [56.50 to 98.01] | 50.0 [9.45 to 90.55] | 100 [34.24 to 100.00] | 75.0 [30.06 to 95.44] | 100 [56.55 to 100.00] | 100 [51.01 to 100.00]

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: Participants who met the following 3 conditions for improvement from baseline of Study M16-063 were classified as meeting the American College of Rheumatology 70% response (ACR70) criteria:
  1. ≥ 70% improvement in 68-tender joint count from Baseline of Study M16-063
  2. ≥ 70% improvement in 66-swollen joint count from Baseline of Study M16-063 and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters from Baseline of Study M16-063:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 10 | 12 | 18 | 8
percentage of participants
  Week 18: number analyzed (Participants) | 23 | 15 | 10 | 12 | 18 | 8
  Week 18 | 47.8 [29.24 to 67.04] | 33.3 [15.18 to 58.29] | 20.0 [5.67 to 50.98] | 25.0 [8.89 to 53.23] | 55.6 [33.72 to 75.44] | 37.5 [13.68 to 69.43]
  Week 24: number analyzed (Participants) | 26 | 14 | 8 | 9 | 16 | 8
  Week 24 | 57.7 [38.95 to 74.46] | 42.9 [21.38 to 67.41] | 12.5 [2.24 to 47.09] | 55.6 [26.67 to 81.12] | 62.5 [38.64 to 81.52] | 87.5 [52.91 to 97.76]
  Week 30: number analyzed (Participants) | 22 | 13 | 7 | 10 | 16 | 8
  Week 30 | 63.6 [42.95 to 80.27] | 46.2 [23.21 to 70.86] | 14.3 [2.57 to 51.31] | 60.0 [31.27 to 83.18] | 68.8 [44.40 to 85.84] | 87.5 [52.91 to 97.76]
  Week 36: number analyzed (Participants) | 23 | 8 | 4 | 9 | 12 | 6
  Week 36 | 78.3 [58.10 to 90.34] | 50.0 [21.52 to 78.48] | 25.0 [4.56 to 69.94] | 44.4 [18.88 to 73.33] | 75.0 [46.77 to 91.11] | 66.7 [30.00 to 90.32]
  Week 48: number analyzed (Participants) | 17 | 6 | 4 | 7 | 8 | 6
  Week 48 | 58.8 [36.01 to 78.39] | 50.0 [18.76 to 81.24] | 25.0 [4.56 to 69.94] | 42.9 [15.82 to 74.95] | 75.0 [40.93 to 92.85] | 83.3 [43.65 to 96.99]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 4 | 5 | 4
  Week 60 | 88.9 [56.50 to 98.01] | 50.0 [9.45 to 90.55] | 50.0 [9.45 to 90.55] | 25.0 [4.56 to 69.94] | 60.0 [23.07 to 88.24] | 75.0 [30.06 to 95.44]

11. Secondary Outcome: Change in Swollen Joint Count 66 (SJC66) From Baseline of Study M16-063
Description: Sixty-six joints were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with swelling) to 66 (worst possible score/66 joints with swelling). Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: swollen joint counts
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 28 | 16 | 11 | 12 | 20 | 9
swollen joint counts
  Week 18 | -11.50 [-13.66 to -9.34] | -9.88 [-14.37 to -5.38] | -8.00 [-11.28 to -4.72] | -13.42 [-18.40 to -8.43] | -12.80 [-16.11 to -9.49] | -9.78 [-13.06 to -6.50]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 8
  Week 24 | -11.67 [-13.85 to -9.49] | -10.54 [-14.25 to -6.82] | -7.67 [-10.13 to -5.21] | -15.60 [-21.14 to -10.06] | -13.24 [-16.48 to -9.99] | -10.38 [-14.22 to -6.53]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | -11.87 [-14.53 to -9.21] | -7.69 [-11.64 to -3.74] | -5.86 [-8.27 to -3.44] | -15.50 [-21.05 to -9.95] | -13.44 [-17.11 to -9.77] | -10.75 [-14.61 to -6.89]
  Week 36: number analyzed (Participants) | 24 | 8 | 4 | 10 | 12 | 6
  Week 36 | -12.38 [-14.84 to -9.91] | -10.13 [-13.42 to -6.83] | -7.75 [-11.73 to -3.77] | -14.60 [-21.38 to -7.82] | -14.25 [-18.71 to -9.79] | -10.50 [-14.79 to -6.21]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 6
  Week 48 | -13.67 [-16.57 to -10.77] | -8.00 [-16.13 to 0.13] | -8.00 [-11.90 to -4.10] | -15.88 [-21.34 to -10.41] | -15.75 [-21.84 to -9.66] | -10.67 [-15.34 to -5.99]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -14.44 [-17.73 to -11.16] | -12.50 [-18.85 to -6.15] | -7.50 [-39.27 to 24.27] | -15.40 [-23.66 to -7.14] | -13.00 [-20.80 to -5.20] | -11.25 [-16.00 to -6.50]

12. Secondary Outcome: Change in Tender Joint Count 68 (TJC68) From Baseline of Study M16-063
Description: Sixty-eight joints were assessed for tenderness by physical examination. Pain or tenderness of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with tenderness) to 68 (worst possible score/68 joints with tenderness). Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: tender joint counts
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 28 | 16 | 11 | 12 | 20 | 9
tender joint counts
  Week 18 | -17.29 [-20.95 to -13.62] | -12.69 [-18.77 to -6.61] | -9.82 [-13.63 to -6.01] | -14.17 [-21.70 to -6.63] | -19.75 [-25.63 to -13.87] | -10.67 [-16.21 to -5.12]
  Week 24: number analyzed (Participants) | 27 | 13 | 9 | 10 | 17 | 8
  Week 24 | -17.93 [-21.84 to -14.02] | -15.77 [-19.37 to -12.17] | -8.11 [-10.95 to -5.28] | -20.20 [-26.97 to -13.43] | -20.76 [-27.39 to -14.14] | -14.25 [-18.44 to -10.06]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | -16.30 [-20.32 to -12.29] | -9.54 [-18.16 to -0.92] | -4.57 [-7.29 to -1.86] | -19.80 [-27.25 to -12.35] | -20.50 [-28.45 to -12.55] | -14.88 [-18.60 to -11.15]
  Week 36: number analyzed (Participants) | 24 | 8 | 4 | 10 | 12 | 6
  Week 36 | -16.42 [-20.15 to -12.68] | -15.25 [-19.85 to -10.65] | -8.00 [-15.46 to -0.54] | -18.40 [-26.99 to -9.81] | -24.92 [-33.96 to -15.88] | -14.83 [-19.21 to -10.46]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 6
  Week 48 | -17.33 [-21.05 to -13.61] | -12.33 [-23.09 to -1.58] | -5.50 [-14.64 to 3.64] | -18.88 [-28.63 to -9.12] | -28.88 [-41.80 to -15.95] | -15.00 [-20.10 to -9.90]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -19.78 [-25.14 to -14.41] | -19.00 [-82.53 to 44.53] | -11.50 [-81.38 to 58.38] | -20.20 [-35.42 to -4.98] | -26.20 [-36.90 to -15.50] | -15.50 [-21.52 to -9.48]

13. Secondary Outcome: Change in Participant's Assessment of Pain (Visual Analog Scale [VAS]) From Baseline of Study M16-063
Description: Participants rated their pain on a visual analogue scale (VAS) of 0 to 100 (mm), with 0 representing no pain and 100 representing the worst possible pain. Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 7 | 10 | 18 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 10 | 18 | 8
  Week 18 | -49.68 [-62.42 to -36.94] | -34.67 [-51.73 to -17.61] | -25.57 [-56.51 to 5.37] | -32.50 [-53.25 to -11.75] | -56.17 [-72.40 to -39.93] | -47.88 [-76.92 to -18.83]
  Week 24: number analyzed (Participants) | 26 | 14 | 7 | 10 | 17 | 8
  Week 24 | -45.46 [-58.31 to -32.61] | -48.36 [-60.60 to -36.11] | -29.43 [-50.47 to -8.39] | -42.00 [-61.74 to -22.26] | -57.76 [-73.67 to -41.86] | -59.38 [-80.35 to -38.40]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 10 | 16 | 8
  Week 30 | -48.18 [-61.90 to -34.46] | -40.62 [-63.40 to -17.83] | -20.00 [-48.48 to 8.48] | -45.90 [-70.64 to -21.16] | -53.63 [-71.19 to -36.06] | -60.25 [-80.74 to -39.76]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 10 | 12 | 6
  Week 36 | -49.22 [-61.84 to -36.59] | -47.13 [-72.05 to -22.20] | -25.67 [-120.27 to 68.94] | -46.70 [-63.40 to -30.00] | -58.83 [-80.69 to -36.98] | -54.83 [-90.68 to -18.98]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 8 | 8 | 6
  Week 48 | -60.06 [-72.78 to -47.34] | -49.00 [-72.85 to -25.15] | -35.00 [-69.15 to -0.85] | -56.13 [-82.80 to -29.45] | -58.75 [-82.80 to -34.70] | -61.50 [-94.46 to -28.54]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -54.67 [-77.99 to -31.34] | -52.00 [-522.13 to 418.13] | -45.50 [-140.80 to 49.80] | -58.80 [-73.74 to -43.86] | -61.00 [-88.13 to -33.87] | -55.00 [-100.36 to -9.64]

14. Secondary Outcome: Change in Patient's Global Assessment of Disease Activity (PtGA) From Baseline of Study M16-063
Description: Participants rated their disease activity for the past 24 hours using a Patient's Global Assessment of Disease Activity Global visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 26 | 15 | 7 | 10 | 18 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 10 | 18 | 8
  Week 18 | -45.18 [-58.36 to -32.00] | -34.07 [-50.11 to -18.03] | -28.57 [-61.69 to 4.55] | -35.70 [-56.96 to -14.44] | -56.56 [-72.18 to -40.93] | -40.13 [-67.21 to -13.04]
  Week 24: number analyzed (Participants) | 26 | 14 | 7 | 10 | 17 | 8
  Week 24 | -48.62 [-59.37 to -37.87] | -45.93 [-60.14 to -31.72] | -33.29 [-59.62 to -6.95] | -45.20 [-61.30 to -29.10] | -62.47 [-76.09 to -48.85] | -58.13 [-74.96 to -41.29]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 10 | 16 | 8
  Week 30 | -46.18 [-60.77 to -31.60] | -39.69 [-61.63 to -17.76] | -21.40 [-57.54 to 14.74] | -45.20 [-67.27 to -23.13] | -56.31 [-71.70 to -40.92] | -57.75 [-75.80 to -39.70]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 10 | 12 | 6
  Week 36 | -51.70 [-64.00 to -39.39] | -48.63 [-73.95 to -23.30] | -31.67 [-141.65 to 78.32] | -46.20 [-64.52 to -27.88] | -61.00 [-81.17 to -40.83] | -53.33 [-84.24 to -22.42]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 8 | 8 | 6
  Week 48 | -54.24 [-69.66 to -38.81] | -44.00 [-71.07 to -16.93] | -38.67 [-88.62 to 11.28] | -53.13 [-76.82 to -29.43] | -60.75 [-84.13 to -37.37] | -56.67 [-84.14 to -29.19]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -56.67 [-83.18 to -30.16] | -56.00 [-462.60 to 350.60] | -54.50 [-226.03 to 117.03] | -54.60 [-70.61 to -38.59] | -59.80 [-96.50 to -23.10] | -57.00 [-87.75 to -26.25]

15. Secondary Outcome: Change in Physician's Global Assessment of Disease Activity (PhGA) From Baseline of Study M16-063
Description: The physician assessed a participant's disease activity at the time of the visit using a Physician's Global Assessment of Disease visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 27 | 15 | 7 | 9 | 17 | 8
units on a scale
  Week 18: number analyzed (Participants) | 23 | 15 | 7 | 7 | 17 | 8
  Week 18 | -57.22 [-65.56 to -48.87] | -41.00 [-53.42 to -28.58] | -33.00 [-61.23 to -4.77] | -35.00 [-59.98 to -10.02] | -59.06 [-69.39 to -48.72] | -55.13 [-82.03 to -28.22]
  Week 24: number analyzed (Participants) | 27 | 14 | 7 | 9 | 16 | 8
  Week 24 | -57.93 [-65.61 to -50.25] | -48.36 [-60.05 to -36.66] | -39.43 [-70.88 to -7.98] | -50.89 [-68.36 to -33.42] | -61.19 [-71.90 to -50.47] | -62.38 [-77.73 to -47.02]
  Week 30: number analyzed (Participants) | 23 | 13 | 5 | 9 | 15 | 8
  Week 30 | -55.04 [-64.27 to -45.82] | -41.23 [-57.85 to -24.61] | -41.80 [-60.33 to -23.27] | -54.78 [-71.11 to -38.45] | -56.20 [-73.22 to -39.18] | -63.50 [-79.15 to -47.85]
  Week 36: number analyzed (Participants) | 22 | 8 | 3 | 9 | 11 | 6
  Week 36 | -57.55 [-66.96 to -48.13] | -53.75 [-70.49 to -37.01] | -60.00 [-112.58 to -7.42] | -54.78 [-73.97 to -35.58] | -68.45 [-81.66 to -55.25] | -65.83 [-89.60 to -42.06]
  Week 48: number analyzed (Participants) | 18 | 6 | 3 | 7 | 8 | 5
  Week 48 | -56.39 [-71.53 to -41.24] | -36.83 [-75.18 to 1.52] | -56.67 [-93.29 to -20.04] | -57.14 [-80.22 to -34.07] | -66.13 [-82.33 to -49.92] | -66.40 [-89.67 to -43.13]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 4 | 5 | 4
  Week 60 | -64.33 [-79.18 to -49.48] | -56.00 [-437.19 to 325.19] | -65.00 [-141.24 to 11.24] | -61.50 [-88.83 to -34.17] | -60.00 [-88.34 to -31.66] | -56.75 [-87.94 to -25.56]

16. Secondary Outcome: Change in Health Assessment Questionnaire Disability Index (HAQ-DI) From Baseline of Study M16-063
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from baseline in the overall score indicates improvement.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 25 | 15 | 7 | 10 | 17 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 10 | 17 | 8
  Week 18 | -0.57 [-0.84 to -0.29] | -0.49 [-0.84 to -0.14] | -0.61 [-1.27 to 0.06] | -0.61 [-1.04 to -0.19] | -0.85 [-1.21 to -0.50] | -0.47 [-0.77 to -0.17]
  Week 24: number analyzed (Participants) | 25 | 14 | 7 | 10 | 16 | 8
  Week 24 | -0.59 [-0.81 to -0.36] | -0.46 [-0.80 to -0.12] | -0.57 [-1.24 to 0.09] | -0.54 [-0.98 to -0.09] | -0.59 [-0.94 to -0.25] | -0.78 [-1.29 to -0.27]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 10 | 15 | 8
  Week 30 | -0.64 [-0.91 to -0.36] | -0.45 [-0.93 to 0.03] | -0.15 [-0.45 to 0.15] | -0.51 [-0.94 to -0.09] | -0.73 [-1.10 to -0.35] | -0.75 [-1.17 to -0.33]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 10 | 11 | 6
  Week 36 | -0.67 [-0.95 to -0.38] | -0.70 [-1.45 to 0.05] | -0.33 [-0.81 to 0.14] | -0.30 [-0.70 to 0.10] | -0.51 [-0.94 to -0.09] | -0.56 [-1.05 to -0.07]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 8 | 8 | 6
  Week 48 | -0.70 [-1.06 to -0.34] | -0.63 [-1.76 to 0.51] | -0.29 [-0.65 to 0.07] | -0.42 [-0.90 to 0.06] | -0.39 [-0.83 to 0.05] | -0.71 [-1.17 to -0.25]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -0.78 [-1.22 to -0.34] | -0.75 [-13.46 to 11.96] | -0.31 [-4.28 to 3.66] | -0.58 [-1.30 to 0.15] | -0.48 [-1.77 to 0.82] | -0.72 [-1.61 to 0.18]

17. Secondary Outcome: Change in High-Sensitivity C-Reactive Protein (Hs-CRP) From Baseline of Study M16-063
Description: C-reactive protein is a blood test marker for inflammation in the body, and levels rise in response to inflammation. A negative change from baseline indicates improvement.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 28 | 16 | 11 | 12 | 20 | 9
mg/L
  Week 18 | -16.04 [-24.13 to -7.95] | 5.34 [-9.84 to 20.53] | -0.96 [-6.20 to 4.28] | -14.85 [-34.27 to 4.57] | -11.48 [-16.88 to -6.07] | -10.00 [-28.36 to 8.35]
  Week 24: number analyzed (Participants) | 27 | 14 | 9 | 10 | 17 | 7
  Week 24 | -15.08 [-23.26 to -6.90] | -0.20 [-15.16 to 14.76] | -2.18 [-4.30 to -0.06] | -15.09 [-38.53 to 8.34] | -9.48 [-15.35 to -3.60] | -13.16 [-32.31 to 5.99]
  Week 30: number analyzed (Participants) | 23 | 13 | 7 | 10 | 16 | 8
  Week 30 | -16.61 [-27.35 to -5.88] | -6.00 [-24.37 to 12.36] | -1.66 [-4.91 to 1.59] | -17.11 [-44.18 to 9.95] | -9.55 [-14.24 to -4.85] | -16.22 [-28.83 to -3.61]
  Week 36: number analyzed (Participants) | 24 | 8 | 4 | 10 | 12 | 6
  Week 36 | -13.88 [-23.43 to -4.32] | -12.43 [-27.58 to 2.73] | -1.58 [-11.33 to 8.18] | -13.61 [-34.50 to 7.28] | -7.76 [-13.95 to -1.56] | -18.34 [-37.30 to 0.62]
  Week 48: number analyzed (Participants) | 18 | 6 | 4 | 8 | 8 | 6
  Week 48 | -16.41 [-28.14 to -4.69] | -18.38 [-50.37 to 13.60] | -5.99 [-17.43 to 5.45] | -20.18 [-49.36 to 9.00] | -7.22 [-14.57 to 0.14] | -18.30 [-36.16 to -0.44]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -25.69 [-45.41 to -5.98] | -31.46 [-288.63 to 225.71] | -3.98 [-116.05 to 108.09] | -25.58 [-67.98 to 16.83] | -3.34 [-23.18 to 16.50] | -12.47 [-33.61 to 8.67]

18. Secondary Outcome: Change in Morning Stiffness Severity From Baseline of Study M16-063
Description: Morning stiffness severity was assessed by a numeric rating-scale (NRS). Participants rated the severity of morning stiffness during the past week from 0 to 10 with 0 representing "not severe" and 10 "very severe". Negative values indicate improvement from baseline.
Time Frame: Baseline in Study M16-063, Weeks 18, 24, 30, 36, 48, and 60 in Study M16-763
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
Number analyzed (Participants) | 25 | 15 | 7 | 10 | 17 | 8
units on a scale
  Week 18: number analyzed (Participants) | 22 | 15 | 7 | 10 | 17 | 8
  Week 18 | -4.27 [-5.56 to -2.99] | -2.27 [-3.69 to -0.84] | -2.14 [-4.99 to 0.70] | -3.40 [-6.02 to -0.78] | -5.29 [-6.54 to -4.05] | -2.38 [-4.65 to -0.10]
  Week 24: number analyzed (Participants) | 25 | 14 | 7 | 10 | 16 | 8
  Week 24 | -4.48 [-5.52 to -3.44] | -2.64 [-3.81 to -1.47] | -3.29 [-5.89 to -0.69] | -3.70 [-5.21 to -2.19] | -4.88 [-6.43 to -3.32] | -3.50 [-5.50 to -1.50]
  Week 30: number analyzed (Participants) | 22 | 13 | 5 | 10 | 15 | 8
  Week 30 | -4.36 [-5.83 to -2.90] | -2.23 [-4.28 to -0.18] | -1.20 [-2.82 to 0.42] | -4.20 [-5.66 to -2.74] | -4.53 [-5.75 to -3.32] | -3.13 [-5.55 to -0.70]
  Week 36: number analyzed (Participants) | 23 | 8 | 3 | 10 | 11 | 6
  Week 36 | -4.43 [-5.95 to -2.92] | -3.38 [-5.74 to -1.01] | -1.00 [-5.30 to 3.30] | -4.00 [-5.39 to -2.61] | -5.55 [-6.80 to -4.29] | -3.00 [-6.18 to 0.18]
  Week 48: number analyzed (Participants) | 17 | 6 | 3 | 8 | 8 | 6
  Week 48 | -5.47 [-6.64 to -4.30] | -3.33 [-6.49 to -0.17] | -1.00 [-7.57 to 5.57] | -4.13 [-6.67 to -1.58] | -5.38 [-7.10 to -3.65] | -3.67 [-6.90 to -0.44]
  Week 60: number analyzed (Participants) | 9 | 2 | 2 | 5 | 5 | 4
  Week 60 | -4.89 [-6.54 to -3.24] | -4.50 [-23.56 to 14.56] | -3.00 [NA to NA] — Not calculable/estimable because standard deviation = 0 | -4.40 [-6.66 to -2.14] | -4.80 [-7.19 to -2.41] | -3.00 [-5.25 to -0.75]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study; median time on follow-up was ABBV-599 in M16-063/M16-763 (279 days); ABBV-105 60 mg/UPA placebo (183 days); ABBV-105 20 mg/UPA placebo (159 days); ABBV-105 5 mg/UPA placebo (337 days); UPA 15 mg/ABBV-105 placebo (229 days); and Placebo in M16-063/ABBV-599 in M16-763 (281 days). TEAEs/SAEs were collected from the first dose in M16-763 until 30 days after last dose, up to 52 weeks.
Description: All-cause mortality and adverse events: all participants who completed Study M16-063 and received at least one dose of assigned study drug in Study M16-763, grouped according to treatments actually received in Study M16-763
Arm/Group | ABBV-599 in M16-063/ABBV-599 in M16-763 | ABBV-105 60 mg/UPA Placebo | ABBV-105 20 mg/UPA Placebo | ABBV-105 5 mg/UPA Placebo | UPA 15 mg/ABBV-105 Placebo | Placebo in M16-063/ABBV-599 in M16-763
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/16 | 0/12 | 0/12 | 0/20 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/16 | 0/12 | 0/12 | 1/20 | 0/9
Other Adverse Events (participants affected / at risk) | 8/28 | 10/16 | 3/12 | 5/12 | 7/20 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-599 in M16-063/ABBV-599 in M16-763 (N=28) | ABBV-105 60 mg/UPA Placebo (N=16) | ABBV-105 20 mg/UPA Placebo (N=12) | ABBV-105 5 mg/UPA Placebo (N=12) | UPA 15 mg/ABBV-105 Placebo (N=20) | Placebo in M16-063/ABBV-599 in M16-763 (N=9)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-599 in M16-063/ABBV-599 in M16-763 (N=28) | ABBV-105 60 mg/UPA Placebo (N=16) | ABBV-105 20 mg/UPA Placebo (N=12) | ABBV-105 5 mg/UPA Placebo (N=12) | UPA 15 mg/ABBV-105 Placebo (N=20) | Placebo in M16-063/ABBV-599 in M16-763 (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG INTOLERANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
URETHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINE ANALYSIS ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL CYST (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03823378/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03823378/SAP_001.pdf